CLINICAL TRIAL: NCT01878838
Title: A Prospective Randomized Controlled Clinical Trial Comparing the Intra-operative Effects, Safety, Efficacy and Performance of Two Commercially Available Laser Systems in Patients Undergoing Femtosecond Laser-Assisted Cataract Surgery.
Brief Title: The Comparison of Cataract Lasers Using the Optimedica Catalys Laser and the Alcon LenSx Laser.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven H. Linn, OD (Other)
Responsible Party: Sponsor-Investigator, Steven H. Linn, OD, Study Coordinator, Hoopes Vision
Organization: Hoopes Vision (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HV-AVO1
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Nuclear Sclerosis of the Lens; Posterior Subcapsular Cataract; Cortical Cataract
MeSH Terms: conditions — Cataract, Age-Related Nuclear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catalys Treated Eyes (Active Comparator): Patient's aged 22 and older with visually significant cataracts undergoing Femtosecond Laser Assisted Cataract Surgery w/ Catalys Laser
  Interventions: Procedure: Femtosecond Laser Assisted Cataract Surgery w/ Catalys Laser
- LenSx Treated Eyes (Active Comparator): Patient's aged 22 and older with visually significant cataracts undergoing Femtosecond Laser Assisted Cataract Surgery w/ LenSx Laser.
  Interventions: Procedure: Femtosecond Laser Assisted Cataract Surgery w/ LenSx Laser

INTERVENTIONS:
Procedure: Femtosecond Laser Assisted Cataract Surgery w/ Catalys Laser — Cohort subjects will undergo Femtosecond Laser Assisted Cataract Surgery in both eyes, with the Optimedica Catalys laser on one eye, and the Alcon LensX laser on the other. First eyes will be randomized.
  Other Names: Optimedica Catalys Precision Laser System
  Arms: Catalys Treated Eyes
Procedure: Femtosecond Laser Assisted Cataract Surgery w/ LenSx Laser — Cohort subjects will undergo Femtosecond Laser Assisted Cataract Surgery in both eyes, with the Optimedica Catalys laser on one eye, and the Alcon LensX laser on the other. First eyes will be randomized.
  Other Names: Alcon LenSx Laser System
  Arms: LenSx Treated Eyes

SUMMARY:
This study compares two FDA approved Cataract Lasers.

DETAILED DESCRIPTION:
The purpose of this study is to systematically evaluate the performance of two commercially available and FDA cleared femtosecond laser systems in patients undergoing femtosecond laser-assisted cataract surgery. Objective data on the repeatability and accuracy of the studied parameters will be gathered and reported as endpoints of the study.

The two systems studied are the Catalys™ Precision Laser System (OptiMedica, CA, USA) and the LenSx® Laser System (Alcon Laboratories, Inc., Fort Worth, TX).

Published data have suggested that the femtosecond laser is a useful tool for cataract surgery.

This study is to determine whether differences or similarities exist in specific treatment parameters achieved with two FDA cleared and commercially available femtosecond laser cataract surgery platforms

ELIGIBILITY:
Inclusion Criteria:

* Have grade 2 to 4 nuclear sclerotic and or cortical or posterior subcapsular cataracts with visual impairment.
* Pupillary dilation of at least 6.0 mm
* Axial length between 21 mm to 26 mm
* Age ≥ 22 years of either gender
* Require laser assisted corneal incisions, capsulotomy and nucleus segmentation
* Understand and sign a written Informed Consent form
* Be able to comply with the treatment and follow-up schedule

Exclusion Criteria:

* Enrolment in another drug or device study within the prior 3 months
* History of ocular trauma
* Acute or chronic disease or illness that would increase risk or confound study results (e.g., uncontrolled diabetes mellitus, immunocompromised, etc.)
* Uncontrolled systemic or ocular disease
* Corneal abnormalities (e.g., stromal, epithelial or endothelial dystrophies, severe corneal opacities, significant corneal edema, etc)
* Diminished aqueous clarity that obscures OCT imaging of the anterior lens capsule
* Corneal ring and/or inlay implant(s)
* Pseudoexfoliation
* Known steroid IOP responder or ocular hypertension IOP >25 mmHg by tonometry
* Retinal detachment within the last 6 months
* Anterior chamber depth less than 2.5 mm

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Dissipated Energy | Intraoperative
  The total amount of phacoemulsification energy delivered during the procedure.

SECONDARY OUTCOMES:
Complete Laser Capsulotomy | Intraoperative
  Did the laser perform a complete capsulotomy with no tags or untreated segments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Rivera, MD, Principal Investigator — Hoopes Vision; Steven H Linn, OD, Study Director — Hoopes Vision
Locations (1):
- Hoopes Vision, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Cullen KA, Hall MJ, Golosinskiy A. Ambulatory surgery in the United States, 2006. Natl Health Stat Report. 2009 Jan 28;(11):1-25. PMID 19294964
- [Background] Vasavada AR, Vasavada V, Vasavada VA, Praveen MR, Johar SR, Gajjar D, Arora AI. Comparison of the effect of torsional and microburst longitudinal ultrasound on clear corneal incisions during phacoemulsification. J Cataract Refract Surg. 2012 May;38(5):833-9. doi: 10.1016/j.jcrs.2011.11.050. PMID 22520307
- [Background] Georgescu D, Kuo AF, Kinard KI, Olson RJ. A fluidics comparison of Alcon Infiniti, Bausch & Lomb Stellaris, and Advanced Medical Optics Signature phacoemulsification machines. Am J Ophthalmol. 2008 Jun;145(6):1014-1017. doi: 10.1016/j.ajo.2008.01.024. Epub 2008 Mar 17. PMID 18343350
- [Background] Dooley IJ, O'Brien PD. Subjective difficulty of each stage of phacoemulsification cataract surgery performed by basic surgical trainees. J Cataract Refract Surg. 2006 Apr;32(4):604-8. doi: 10.1016/j.jcrs.2006.01.045. PMID 16698480
- [Background] Gimbel HV, Neuhann T. Development, advantages, and methods of the continuous circular capsulorhexis technique. J Cataract Refract Surg. 1990 Jan;16(1):31-7. doi: 10.1016/s0886-3350(13)80870-x. PMID 2299571
- [Background] Friedman NJ, Palanker DV, Schuele G, Andersen D, Marcellino G, Seibel BS, Batlle J, Feliz R, Talamo JH, Blumenkranz MS, Culbertson WW. Femtosecond laser capsulotomy. J Cataract Refract Surg. 2011 Jul;37(7):1189-98. doi: 10.1016/j.jcrs.2011.04.022. PMID 21700099
- [Background] Artzen D, Lundstrom M, Behndig A, Stenevi U, Lydahl E, Montan P. Capsule complication during cataract surgery: Case-control study of preoperative and intraoperative risk factors: Swedish Capsule Rupture Study Group report 2. J Cataract Refract Surg. 2009 Oct;35(10):1688-93. doi: 10.1016/j.jcrs.2009.05.026. PMID 19781460
- [Background] Bellini LP, Brum GS, Grossi RS, Borowsky C. Cataract surgery complication rates. Ophthalmology. 2008 Aug;115(8):1432; author reply 1432-3. doi: 10.1016/j.ophtha.2008.04.009. No abstract available. PMID 18675698
- [Background] Richard J, Hoffart L, Chavane F, Ridings B, Conrath J. Corneal endothelial cell loss after cataract extraction by using ultrasound phacoemulsification versus a fluid-based system. Cornea. 2008 Jan;27(1):17-21. doi: 10.1097/ICO.0b013e3181583115. PMID 18245961
- [Background] Hayashi K, Hayashi H, Nakao F, Hayashi F. Risk factors for corneal endothelial injury during phacoemulsification. J Cataract Refract Surg. 1996 Oct;22(8):1079-84. doi: 10.1016/s0886-3350(96)80121-0. PMID 8915805
- [Background] Uy HS, Edwards K, Curtis N. Femtosecond phacoemulsification: the business and the medicine. Curr Opin Ophthalmol. 2012 Jan;23(1):33-9. doi: 10.1097/ICU.0b013e32834cd622. PMID 22081031